CLINICAL TRIAL: NCT04107350
Title: The Whole Body Vibration Training for Total Knee arthroplasty-the Improvement of the Lower Limb
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KMUHIRB-F(II)-20170135
Record Dates: First submitted 2019-09-16; First posted 2019-09-27 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2018-03

CONDITIONS: Knee Osteoarthritis; Arthroplasty Complications; Swelling; Leg
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: knee osteoarthritis status post total knee arthroplasty receive therapy on post-operation day 2 and post operation day 3 Study group: WBV+conventional physical therapy Control group: convention physical therapy
Who Masked: Participant
Masking Description: A single-blinded randomized control trial Intervention by the physical therapist Evaluation by the physician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- whole body vibration on (Experimental): vibration machine on combined with conventional physical therapy
  Interventions: Device: whole-body vibration
- whole body vibration off (Sham Comparator): vibration machine off combined with conventional physical therapy
  Interventions: Device: whole-body vibration

INTERVENTIONS:
Device: whole-body vibration — 10 minutes WBV exercise in standing position; amplitude 2mm,; frequency 4-10Hz; resting interval: 3 minutes rest.

SUMMARY:
Knee Osteoarthritis in elder cause pain and decrease their functional activity. After conservative rehabilitation failure, they might receive total knee arthroplasty. The post-operation rehabilitation could improve range of motion and might help them to back activities of daily Living earlier. However, the pain and swelling after the operation of total knee arthroplasty cause the limitation of early mobilization, cause ROM limitation, muscle strength decrease, functional activity decrease, and impaired activity of daily life. In recent studies, the effect of whole body vibration included improving pain, swelling, muscle strength, balance, and functional activity, increasing metabolic rate and decreasing lactate accumulation. the investigators expect the early intervention of whole body vibration and traditional physical therapy on the post-TKA patient could improve ROM, decrease swelling, increased muscle strength, functional activity, and balance as compared with traditional physical therapy.

DETAILED DESCRIPTION:
1. Name: whole body vibration BW-750
2. Dosage form: frequency 4-10 Hz, 10-15minutes with rest for 3-5 minutes * 2 days in standing position
3. Dose(s): post-op day2, WBV 4-10 Hz, 10-15minutes with rest for 3-5 minutes, post-op day3 WBV 4-10 Hz, 10-15 minutes with 3-5 minutes in standing position
4. Dosing schedule: whole body vibration 4-10 Hz for 10-15 minutes with rest 3-5 minutes on post-op day 2 and day3
5. Mechanism of action: passive muscle contraction, improve swelling, increase blood flow, and improve muscle strength
6. Pharmacological category: N/A

IV.Study design 1. ■ Control: ■ placebo 2. Blinding: ■ double blind 3. Randomized: ■ yes □ no 4. ■ Parallel 5. Duration of study:from IRB approval ~to 31 , Dec. , 2019 6. Number of subjects: 52 persons 7. Is there any of the followings included DSMB, Data Safety Monitoring Board:

* no V.Assessment criteria 1. Efficacy: pain (VAS)，swelling circumference，knee range of motion，knee extensor muscle strength，time up and go，and Activities of Daily Living 2. Safety: The duration and frequency of whole body vibration is relative low. The risk of damage is very low 3. Pharmacokinetics: Not apply 4. Quality of life: Through facilitate muscle contraction, improve blood flow, and decrease pain could improve muscle power, increase range of motion and ADL VI. Selection criteria

  1. Main inclusion criteria: knee osteoarthritis, post-operation of total knee arthroplasty, single leg
  2. Main exclusion criteria: vital signs unstable, uncontrolled blood pressure, diabetes mellitus, neoplasm, neurological disorder, fibromyalgia, cardiac pacemaker, bilateral TKA, musculoskeletal involvement other than TKA VII.Study procedures(summary)

  <!-- -->

  1. Written informed consent must be obtained before any study specific procedures are undertaken.
  2. The process of the experiment (brief describe)

  <!-- -->

  1. Randomized distribute participants into two groups, "whole body vibration(experimental group)+ traditional physical therapy" group and "placebo group with traditional physical therapy+ whole body vibration (placebo without turn-on vibration)".
  2. Post-TKA day 1 (not op day) Pre-test (baselin data) include pain(VAS), leg circumference, knee ROM, knee extensor strength (JAMMAR), sit to stand average duration, 6 meters ambulatory test.

     Both groups receive traditional physical therapy and passive continuous passive motion (CPM).
  3. Post-TKA day 2 Both groups keep traditional physical therapy and CPM.

  (1) The experimental group perform pre-test before the treatment. After the pre-test, participants receive 10-15 minutes WBV exercise in standing position, amplitude 2mm, frequency 4-10Hz, with rest about 3-5minutes. After the treatment, perform post-treatment test 1.

  (2) The control group standing on the WBV machine without turn-on for 10-15 minutes and then post-treatment test 1.

  4. Post-TKA day 3
  1. The experimental group participants receive 10-15 minutes WBV exercise in standing position, amplitude 2mm, frequency 4-10 Hz, with rest about 3-5minutes. After the treatment, perform post-treatment test 2.
  2. The control group standing on the WBV machine without turn-on for 10-15 minutes and then post-treatment test 1.

     Statistical analysis 1. Statistical Method for Efficacy / Safety measurements: Demographic data were collected on age, pre-TKA Osteoarthritis X-ray Kellgren-Lawrence classification, sex, weight, height, side of involvement. The investigators use t-test, or chi-square test to confirm homogeneity.

     On the other side, measurement the circulation of the affected limb above knee 15 cm, knee and below knee 5cm for swelling evaluation. Pain scale with Numeric Rating Scale; NRS) before intervention, post-test 1 and post-test 2. Muscle power of knee extensor by the duration with holding knee extension in sitting position before intervention, post-test 1 and post-test 2 Knee range of motion with goniometer in sitting (prone position) The duration of time up and go，6 meter ambulation test with walker usage. ADL evaluation with Barthel Index including transfer score, ambulation score, and up/down stairs score. Paired t-test is applied for statistical significance between these measurements.

     Discussion The investigator expected that post treatment, the patients in the vibration group got increases in knee extensor strength, improvement in calf swelling and functional performance when compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* knee osteoarthritis
* post-operation of total knee arthroplasty
* single leg knee arthroplasty

Exclusion Criteria:

* vital signs unstable
* uncontrolled blood pressure
* diabetes mellitus
* neoplasm
* neurological disorder
* fibromyalgia
* cardiac pacemaker
* musculoskeletal involvement other than TKA

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
pain scale (Numeric Rating Scale 0-10) | 30 seconds
  pain with NRS before and after therapy
lower leg circumference (cm) | 1 minute
  Above knee 15cm and below knee 5cm circumference before and after therapy
knee range of motion | 30 seconds
  knee range of motion in degree with goniometer in supine position
knee extensor muscle strength | 1 minute
  knee extensor strength with dynamometer in knee flexion 45 degree, in kg in 3 times

SECONDARY OUTCOMES:
Modified five times sit to stand test | 5 minutes
  straight back chair with a solid seat 40 cm high. The investigator asked the participants to stand up and sit down as quickly as possible for 5 times, and the time spent were recorded.
Modified timed up and go (TUG) test | 5 minutes
  stand from seat height of 40 cm, walk a distance of 3 meters, turn around, walk back to the chair and sit down

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hsin Chen, PhD, Study Chair — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park YG, Kwon BS, Park JW, Cha DY, Nam KY, Sim KB, Chang J, Lee HJ. Therapeutic effect of whole body vibration on chronic knee osteoarthritis. Ann Rehabil Med. 2013 Aug;37(4):505-15. doi: 10.5535/arm.2013.37.4.505. Epub 2013 Aug 26. PMID 24020031

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-14): https://cdn.clinicaltrials.gov/large-docs/50/NCT04107350/Prot_SAP_000.pdf